CLINICAL TRIAL: NCT03776760
Title: Strategies for Hepatitis C Testing and Treatment in Aboriginal Communities That Lead to Elimination
Acronym: SCALE-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kirby Institute (Other Government)
Collaborators: South Australian Health and Medical Research Institute (Other); Flinders University (Other)
Responsible Party: Sponsor
Other Study IDs: VHCRP1802
Record Dates: First submitted 2018-11-21; First posted 2018-12-17 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis C; Hepatitis; Liver Diseases; Hepatitis, Viral, Human; RNA Virus Infections; Digestive System Diseases
MeSH Terms: conditions — Hepatitis C; Hepatitis; Liver Diseases; Hepatitis, Viral, Human; RNA Virus Infections; Digestive System Diseases | interventions — Sofosbuvir; sofosbuvir-velpatasvir drug combination; glecaprevir and pibrentasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried Blood Spot samples for HCV RNA viral load testing and viral genome sequencing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fingerstick Point of Care GeneXpert HCV Test: Participants will have HCV testing using the finger-stick point of care GeneXpert quantitative HCV RNA assay.
  Interventions: Device: Fingerstick GeneXpert HCV RNA quantitative assay; Drug: sofosbuvir/velpatesvir; Drug: glecaprevir/pibrentasvir
- Treat - SOF/VEL: Participants with active HCV infection will be offered treatment with one of two pan-genoptyic regimens available in Australia - sofosbuvir/velpatesvir
  Interventions: Drug: sofosbuvir/velpatesvir
- Treat - G/P: Participants with active HCV infection will be offered treatment with one of two pan-genoptyic regimens available in Australia - glecaprevir/pibrentasvir
  Interventions: Drug: glecaprevir/pibrentasvir

INTERVENTIONS:
Device: Fingerstick GeneXpert HCV RNA quantitative assay — All participants at risk of HCV infection will receive HCV RNA testing using the GeneXpert finger-stick point-of-care HCV quantitative assay 6 monthly
  Groups: Fingerstick Point of Care GeneXpert HCV Test
Drug: sofosbuvir/velpatesvir — Participants with active HCV infection will be offered treatment with one of two pan-genotypic regimens available in Australia
  Other Names: Epclusa
  Groups: Fingerstick Point of Care GeneXpert HCV Test; Treat - SOF/VEL
Drug: glecaprevir/pibrentasvir — Participants with active HCV infection will be offered treatment with one of two pan-genotypic regimens available in Australia
  Other Names: Maviret
  Groups: Fingerstick Point of Care GeneXpert HCV Test; Treat - G/P

SUMMARY:
A community-based "test and treat" intervention integrating point-of-care HCV RNA testing, non-invasive liver disease assessment and linkage to care will lead to a reduction in HCV prevalence among people attending Aboriginal health services.

DETAILED DESCRIPTION:
SCALE-C is an interventional cohort study recruiting people with or at risk of HCV infection from Aboriginal health services in Australia. Participants will be screened for HCV infection using point-of-care testing (anti-HCV antibody and/or HCV RNA). People with current HCV infection (HCV RNA positive) will be offered treatment with eight or 12 weeks of pan-genotypic DAA therapy, glecaprevir/pibrentasvir or sofosbuvir/velpatasvir, as available on the PBS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* voluntarily signed the informed consent form.

Exclusion Criteria:

* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People attending Aboriginal health services will be invited to receive HCV RNA testing using the GeneXpert fingerstick HCV RNA assay. Those found to have active HCV infection will be offered treatment with one of two pan-genotypic direct acting antiviral therapies available in Australia (SOF/VEL or G/P)
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in Hepatitis C prevalence | Week 0 to week 144
  Change in the proportion of people with current HCV infection (HCV RNA positive)

SECONDARY OUTCOMES:
Change in Hepatitis C incidence | Week 0 to week 144
  Change in HCV incidence will be calculated using person-time of observation.
DAA uptake | To week 144
  Proportion with HCV infection initiating DAA therapy
Treatment response rate (SVR12 rate) | From week 0 to Week 144
  Overall SVR12 rate in those who commence treatment
HCV reinfection incidence post treatment | 6 monthly from end of treatment until week 144
  Participants will be assessed six monthly post end of treatment for HCV recurrence.

OTHER OUTCOMES:
HCV Transmission networks within the Aboriginal community | At screening for all participants
  HCV viral genome for will be sequenced for all participants from their screening sample. The sequences ill be used for develop a phylogenetic tree which can be used to determine transmission networks within the study population.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Jullums Lismore Aboriginal Medical Service, Lismore, New South Wales
  - Walhallow Aboriginal Corporation, Quirindi, New South Wales
  - Pangula Mannamurna Aboriginal Corporation, Mount Gambier, South Australia
  - Port Lincoln Aboriginal Health Service, Port Lincoln, South Australia

REFERENCES:
- [Derived] Hosseini-Hooshyar S, Valerio H, Flynn E, Sexton C, Barzi F, Amarasena S, De Koster L, Sellen D, Winterfield N, Grebely J, Matthews GV, Boyd MA, Applegate TL, Petoumenos K, Lafferty L, Dore GJ, Treloar C, Martinello M, Ward J. A point-of-care testing intervention to improve hepatitis C diagnosis and treatment uptake among people attending Aboriginal community controlled health services: the SCALE-C study. BMC Infect Dis. 2025 Nov 17;25(1):1604. doi: 10.1186/s12879-025-12004-z. PMID 41250046